CLINICAL TRIAL: NCT02953197
Title: 18F-FDG-PET Guided Dose-Painting With Intensity Modulated Radiotherapy in Oropharyngeal Tumours (FiGaRO), A Phase 1 Pilot Study
Brief Title: 18F-FDG-PET Guided Dose-Painting With Intensity Modulated Radiotherapy in Oropharyngeal Tumours
Acronym: FiGaRO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Velindre NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ113/N033
Record Dates: First submitted 2016-10-25; First posted 2016-11-02 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm radiotherapy dose escalation (Experimental): FDG-PET guided radiation dose escalation Selective dose escalation
  Interventions: Radiation: FDG-PET guided radiation dose escalation

INTERVENTIONS:
Radiation: FDG-PET guided radiation dose escalation — Selective dose escalation

SUMMARY:
Treatment of cancers of the head and neck, including oropharyngeal tumours, usually consist of a combination of radiotherapy and chemotherapy, although surgery may also play a part. Radiotherapy works by using the high energy x-rays to destroy cancer cells. Head and neck cancers often respond well to radiotherapy in the first instance and a proportion of patients will be cured by this treatment. However, not all of the cancer cells are destroyed by the combination of radiotherapy and chemotherapy and, in some patients, the cancer does come back.

Studies have suggested that more efficient killing of cancer cells, and therefore, better cure rates, can be achieved by increasing the radiotherapy dose. However, in the past, this was not possible due to side effects. Intensity Modulated Radiotherapy (IMRT) is a new radiotherapy delivery technique that allows better shaping of the dose to the areas that need irradiating with the potential for fewer side effects. If the investigators use IMRT to deliver an intentionally higher dose of radiation (called a boost) to small selected areas whilst, at the same time giving standard treatment doses to the remaining areas, this approach is called IMRT dose-painting. These selected areas can be identified by a scan called 18F-FDG-PET (18F-fluorodeoxyglucose-positron emission tomography, also known as a 'PET' scan) which is a type of scan that can give information about the activity of a cancer.

The purpose of this study is to find out whether the investigators can use IMRT dose-painting to boost the dose to the region inside a tumour which appears most active on 18F-FDG-PET. If this study shows that this approach is well-tolerated, then the investigators may be able to improve cure rates with this treatment. This would need to be tested in a subsequent study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma (SCC) of the oropharynx assessed as either HPV negative or HPV positive with greater than 10 pack year smoking history and N stage at least N2b, to be treated with primary radical neoadjuvant chemotherapy followed by chemo-intensity modulated radiotherapy (chemo-IMRT) to the primary and bilateral neck nodes
* Age ≥ 18 years.
* ≥T2 tumours.
* Staging 18F-FDG-PET/CT showing adequate uptake at the level of the primary tumour.
* WHO performance status 0-2.
* Renal function adequate for cisplatin chemotherapy.
* All patients must be suitable to attend regular follow-up.
* Written informed consent must be obtained in all patients.

Exclusion Criteria:

* Previous radiotherapy to the head and neck region interfering with the protocol treatment plan.
* Previous malignancy except non-melanoma skin cancer.
* Previous or concurrent illness, which in the investigators opinion, would interfere with either completion of therapy or follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-02; Primary Completion 2018-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients suffering grade 3 or more late mucosal toxicity, assessed using the RTOG /EORTC and modified LENTSOMA scale, at one year post treatment | 1 year following completion of treatment in the last study participant

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Guerrero Urbano, Principal Investigator — Guy's & St Thomas' NHS Foundation Trust, London, UK
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michaelidou A, Adjogatse D, Suh Y, Pike L, Thomas C, Woodley O, Rackely T, Palaniappan N, Jayaprakasam V, Sanchez-Nieto B, Evans M, Barrington S, Lei M, Guerrero Urbano T. 18F-FDG-PET in guided dose-painting with intensity modulated radiotherapy in oropharyngeal tumours: A phase I study (FiGaRO). Radiother Oncol. 2021 Feb;155:261-268. doi: 10.1016/j.radonc.2020.10.039. Epub 2020 Nov 5. PMID 33161013